CLINICAL TRIAL: NCT03765359
Title: Metformin Use to Improve Pregnancy Outcome in Women With Type 1 Diabetes. A Randomized Double-blind Placebo-controlled Multicenter Study.
Brief Title: Metformin Use to Improve Pregnancy Outcome in Women With Type 1 Diabetes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Oulu University Hospital (Other); Helsinki University Central Hospital (Other); Central Finland Hospital District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Diabetes2017; 2016-005031-32 (EudraCT Number)
Record Dates: First submitted 2018-04-24; First posted 2018-12-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Pregnancy; Insulin Resistance; Type1diabetes
Keywords: insulin need; diabetic pregnancy; insulin resistance; metformin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: placebo controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metforminhydrochloride (Active Comparator): Metformin medication starts on 12-14 weeks of gestation. The starting dosage is 1 tablet (500 mg) x1 and it is increased gradually 1 tablet a week up to 2+2 tablets (2000mg) daily. Duration of the treatment is approximately until one week before delivery. Otherwise metformin treatment combined with regular insulin and follow-up during pregnancy follows the national guidelines.
  Interventions: Drug: metforminhydrochloride
- Placebo Oral Tablet (Placebo Comparator): Placebo tablets starts on 12-14 weeks of gestation. The starting dosage is 1 tablet x1 and it is increased gradually 1 tablet a week up to 2+2 tablets daily. Duration of the treatment is approximately until one week before delivery. Otherwise placebo treatment combined with regular insulin and follow-up during pregnancy follows the national guidelines.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: metforminhydrochloride — metformin 500 mg tablets and insulin
  Other Names: A10BA02; Diformin; Metformin
  Arms: metforminhydrochloride
Drug: Placebo Oral Tablet — Placebo tablets mimic metformin 500 mg tablets and insulin
  Arms: Placebo Oral Tablet

SUMMARY:
The study investigates whether additional metformin medication in combination with regular insulin treatment will decrease the need of insulin for women with diabetes mellitus type 1 during pregnancy.

DETAILED DESCRIPTION:
Insulin resistance during pregnancy of diabetes mellitus type 1 patients (DM1) increases the need for insulin and makes it more difficult to maintain normoglycemia. Fetal exposure to hyperglycemia induces macrosomia which increases fetal and neonatal morbidity and mortality. Further more obesity and excess weight gain during pregnancy enhances insulin resistance and it's an independent risk factor for fetal macrosomia.

Metformin is a medical treatment for type 2 diabetes (DM2) where consequential pathophysiology includes insulin resistance. It reduces hepatic glucose production and enhances the use of glucose in muscles relieving insulin resistance. Metformin has also found to inhibit weight gain effectively.

Metformin has approved to be safe and effective in patients with gestational diabetes (GDM). It has found to reduce weight gain and improve postprandial blood glucose levels during pregnancy and reduce neonatal birth trauma in GDM. However, there are no previous studies about the use of metformin in pregnant women with DM1.

Two hundred women with DM1 will be randomized to get placebo or metformin in addition to regular insulin treatment. The sample size has been estimated to demonstrate the difference of 15 % in the need to increase insulin dosages during the pregnancy between the study groups.

ELIGIBILITY:
Inclusion Criteria:

* a pregnancy of a woman with type 1 diabetes.

Exclusion Criteria:

* multiple pregnancy, significant underlying disease (hearth disease, kidney transplant, IBD (inflammatory bowel disease ), SLE (systemic lupus erythematosus ), diseases with use of high dosage corticosteroids (severe asthma or rheumatic disease), severe complications of diabetes (nephropathy, neuropathy, gastroparesis or severe retinopathy), substance abuse, smoking, BMI <18, strong early pregnancy nausea (=hyperemesis)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Study is done during pregnancy
Enrollment: 101 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Changes in the insulin need during pregnancy | from 5-10 gestational weeks until the delivery
  The insulin dosage (IU/ml) in two weeks sets

SECONDARY OUTCOMES:
Blood glucose balance during pregnancy HbA1c | from gestational weeks 5 until the delivery
  HbA1c (mmol/mol)
Blood glucose balance during pregnancy AVG, SD, CV | from gestational weeks 5 until the delivery
  mean blood glucose (mmol/l) level, standard deviation (SD) and the coefficient of variation of the blood glucose levels
Change in the weight | from gestational weeks 5 until the delivery
  Weight gain (g) during pregnancy
Change in the blood pressure | from gestational weeks 5 until the delivery
  Blood pressure (mmHg)
Incidence of pre-eclampsia | from gestational weeks 20 until the delivery
  Incidence of pre-eclampsia (%)
Incidence hepatogestosis | from gestational weeks 20 until the delivery
  Incidence hepatogestosis (%)
Pregnancy complications | from gestational weeks 5 until the delivery
  Incidence proteinuria (mg/mmol or mg/d)
macrosomia | from gestational weeks 20 until the delivery
  estimated fetal weight in ultrasound (grams)
Pregnancy complications | 12-22 weeks of gestation
  incidence of miscarriage (intrauterine death before 22 weeks of gestation or fetal weigth under 500g) (%)
Pregnancy complications | 22-40 weeks of gestation
  incidence of intrauterine death (intrauterine death after 22 weeks of gestation or fetal weigth over 500g) (%)
Thigh fractional volume ultrasound | from gestational weeks 20 until delivery
  Fetal weight estimation (g) is specified by thigh fractional volume ultrasound program
Rate of the caesarean sections | The delivery
  Rate of the caesarean sections (%)
Labour | The delivery
  rate of spontaneous delivery (%)
Rate of the operative vaginal deliveries | The delivery
  Rate of the operative vaginal deliveries (%)
Rate of the shoulder dystocia | The delivery
  Rate of the shoulder dystocia (%)
Labor complications | The delivery
  rate of induced delivery (%)
Rate of the perineal tears | The delivery
  Rate of the perineal tears (%)
Postpartum bleeding | The delivery
  postpartum bleeding (ml)
Newborn variables (gestational age) | After the delivery
  Rate of the premature deliveries (=deliveries before 37 weeks of gestation) (%)
Newborn variables | After the delivery
  weight of the newborn (g)
Newborn outcome | After the delivery
  Acidosis of the newborn (pH)
Newborn outcome (intensive care) | After the delivery
  The need of NICU (neonatal intensive care unit) treatment (days)
Newborn outcome (hypoglycemia) | After the delivery
  The occurrence of hypoglycemia (=plasma glucose under 2.6mmol/l or usage of iv glucose infusion) (%)
Newborn outcome (Erb's) | After the delivery
  Incidence of the Erb's paresis (%)
Cost benefit calculations (sick leaves) | from gestational weeks 12 until delivery
  The need of sick leaves during pregnancy (days)
Cost benefit calculations (visits to maternity outpatient clinic or internal medicine policlinic) | 14-40 weeks of gestation
  The need of polyclinical controls during pregnancy (number of visits/pregnancy)
Cost benefit calculations (hospitalization) | 14-40 weeks of gestation
  The need of hospitalization during pregnancy (days/pregnancy)
Cost benefit calculations (all outpatient visits after delivery ) | One year after the delivery
  The need of policlinical controls of the diabetic mother after the delivery (number of visits)
Cost benefit calculations (hospitalization after delivery, all departments) | Up to one year after the delivery
  The need of hospitalization of the diabetic mother after the delivery (days)
Cost benefit calculations (all hospitalization of the child) | Until the age of one year
  The need of hospitalization of the child (days)
Cost benefit calculations (all policlinical controls of the child) | Until the age of one year
  The need of policlinical controls of the child (number of visits)
high sensitive-CRP | 7-10, 26-28 and 34-36 weeks of gestation
  high sensitive-CRP (mg/l)
lipids | 7-10, 26-28 and 34-36 weeks of gestation
  cholesterol, high density lipoprotein, low density lipoprotein, triglyserids (mmol/l)
Inflammatory markers | 7-10, 26-28 and 34-36 weeks of gestation
  adiponectin, leptin, resistin, IL-6, TNF-α (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Kati Tihtonen, PhD, Principal Investigator — Tampere University Hospital, Tampere University
Locations (5):
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Central Finland Health Care District, Jyväskylä
  - Oulu University hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juuma E, Tihtonen K, Metso SE, Hannula PM, Helminen M, Tertti K, Immonen H, Georgiadis L, Vayrynen K, Ahtiainen P, Nikkinen H, Koivikko M, Laivuori H, Uotila J. The Effect of Metformin on Insulin Requirement, Glycaemic Control and Weight Gain in Type 1 Diabetes During Pregnancy-a Randomised, Placebo-Controlled Multicentre Study. Diabetes Metab Res Rev. 2025 Sep;41(6):e70085. doi: 10.1002/dmrr.70085. PMID 40916351